CLINICAL TRIAL: NCT04453345
Title: The Efficacy of Thalidomide Plus Prednisone and Methotrexate for the Symptomatic Large Granular Lymphocytic Leukemia - a Prospective Multicenter Clinical Trial From China
Brief Title: TPM Regimen (Thalidomide, Prednisone and Methotrexate) in LGLL
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: The First Affiliated Hospital of Nanchang University (Other); First Affiliated Hospital of Guangxi Medical University (Other); Henan Cancer Hospital (Other Government); The First Hospital of Jilin University (Other); Central South University (Other); Tianjin First Central Hospital (Other)
Responsible Party: Principal Investigator, Yi Shuhua, principal investigator, Institute of Hematology & Blood Diseases Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2020003-EC-1
Record Dates: First submitted 2020-06-24; First posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: T-LGL Leukemia; Clpd-Nk
Keywords: Large granular lymphocyte leukemia; thalidomide; methotrexate
MeSH Terms: conditions — Leukemia, Large Granular Lymphocytic | interventions — Thalidomide; Prednisone; Methotrexate

STUDY DESIGN:
Intervention Model Description: TPM treatment plan: thalidomide 50-100mg qn + prednisone 0.5-1mg / kg qod +methotrexate 10mg / m2 / week.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TPM regimen (Experimental): thalidomide 50-100mg daily at bedtime + prednisone 0.5mg/kg qod to 1mg/kg qd + methotrexate 10mg/m2 per week. 4 months one cycle, up to 3 cycles. After get partial remission, thalidomide maintenance will continue up to 2 years.
  Interventions: Drug: thalidomide + prednisone + methotrexate

INTERVENTIONS:
Drug: thalidomide + prednisone + methotrexate — thalidomide 50-100mg daily at bedtime + prednisone 0.5mg/kg qod to 1mg/kg qd + methotrexate 10mg/m2 per week. 4 months one cycle, up to 3 cycles. After get partial remission, thalidomide maintenance will continue up to 2 years.
  Other Names: TPM regimen

SUMMARY:
Large granular lymphocytic leukemia (LGLL) is a lymphoproliferative disease, with LGL infiltration in peripheral blood and bone marrow, hepatosplenomegaly, and cytopenia. Both T-LGLL and CLPD-NK are indolent disease and share similar biology and clinical course, and treated under the same strategy. So the investigators put them together as LGLL. The investigators used TPM regimen (thalidomide + prednison + methotrexate ) to treat LGLL since 2013, and 18/20 patients (90%) obtained clinical response, including 80% complete response. Adverse events (AE) of grade 3 and above are rare and safe. Therefore, the investigators designed this multicenter clinical trial to validate the efficacy of the TPM regimen in symptomatic T-LGLL and CLPD-NK.

DETAILED DESCRIPTION:
Because LGLL has continuously activated cytotoxic T lymphocytes, immunosuppressive therapy is the standard first-line therapy for T-LGLL and CLPD-NK. Previous studies showed that the overall response rate (ORR) of first-line oral immunosuppressants ranged from 21% to 85% (median: 50%). Both methotrexate and cyclosporine A are LGLL first-line treatment options, but the CR rate of methotrexate is only 21%, while the CR rate of CsA is less than 5%. There is insufficient evidence for the treatment of LGLL with prednisone and other glucocorticoids, but it can reduce RA-related inflammation and increase granulocyte levels. The TPM regimen was designed by the investigators. A pilot prospect observation showed that 18/20 (90%) patients obtained response, including 80% CR. This study is a prospective multiple center clinical trail to evaluate the efficacy of TPM regimen in the treatment of symptomatic LGLL. Eligible patients choose the initial treatment plan: thalidomide 50-100mg qn+ prednisone 0.5-1mg / kg qod +methotrexate 10mg / m2 / week. Four months is one course. Maximum three courses will be given if there is a response and thalidomide maintenance will be for another year.

ELIGIBILITY:
Inclusion Criteria:

1. The gender of the patient is not limited, and the age is ≥18 years old;
2. Must meet diagnostic criteria of T-LGLL or CLPD-NK according to WHO 2016 version;
3. The patient is treatment naive or received single methotrexate less than 4 weeks and without response. If relapsed or refractory patients, the patients must be naive for both thalidomide and methotrexate.
4. With LGLL treatment indications, it mainly includes (meets at least one of the following conditions):

   1. ANC <0.5 × 10^9 / L
   2. HGB <100g / L or need red blood cell infusion to maintain
   3. PLT <50 × 10^9 / L
   4. Combining autoimmune diseases that require treatment
   5. symptomatic splenomegaly
   6. Severe B symptoms
   7. Pulmonary hypertension.
5. ECOG performance status score is 0-2;
6. The patient's expected survival time is ≥ 6 months.

Exclusion Criteria:

1. Unable to understand or follow the research procedure;
2. Co-occurrent malignant tumors that has to be treated or course the symptom;
3. Other serious diseases, such as liver, kidney, heart, lung, nerve or metabolic diseases, may impede the ability of patients to tolerate methotrexate, cyclophosphamide or cyclosporin A;
4. ALAT / ASAT or alkaline phosphatase> 3 times the normal value;
5. Creatinine clearance <60ml / min;
6. Serological evidence of active infection of HIV, hepatitis C or hepatitis B;
7. Ineffective contraception;
8. Positive pregnancy test;
9. Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2013-05-20 (Actual); Primary Completion 2023-05-20 (Estimated); Study Completion 2025-05-20 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) rate of TPM regimen | From date of TPM treatment until the date of complete response, assessed up to 100 months
  Hb> 120g / L，platelet> 100×109 / L，ANC > 1.5×109 / L），ALC< 4×109 / L，peripheral LGL in normal（< 0.5×109 / L）

SECONDARY OUTCOMES:
Overall response (PR) | From date of TPM treatment until the date of at least partial response, assessed up to 100 months
  improvement in blood counts (ANC > 0.5 × 10^9/L; HGB increased by >1 g/dL; PLT > 50 × 10^9/L), and the absence of required transfusions.
Progression-free survival (PFS) | From date of TPM treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  the length of time during and after the treatment of LGLL
Duration of response (DoR) | From date of getting response until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  the time from response to progression/death (P/D)
overall survival | From date of TPM treatment until the date of death from any cause, assessed up to 180 months
  the length of the patients survival time

CONTACTS AND LOCATIONS:
Overall Officials: Lugui Qiu, Study Director — Blood Disease Hospital, CAMS and Peking Union Medical College
Locations (9):
- China (9):
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji hopital, Huazhong University of Science and Technology, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Affiliated Hospital of Jilin University, Ch’ang-ch’un, Jilin
  - Xijing Hospital, Air Force Military Medical University, Xi’an, Shanxi
  - Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality
  - Tianjin First Central Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dinmohamed AG, Brink M, Visser O, Jongen-Lavrencic M. Population-based analyses among 184 patients diagnosed with large granular lymphocyte leukemia in the Netherlands between 2001 and 2013. Leukemia. 2016 Jun;30(6):1449-51. doi: 10.1038/leu.2016.68. Epub 2016 Apr 8. No abstract available. PMID 27055870
- [Background] Matutes E. Large granular lymphocytic leukemia. Current diagnostic and therapeutic approaches and novel treatment options. Expert Rev Hematol. 2017 Mar;10(3):251-258. doi: 10.1080/17474086.2017.1284585. Epub 2017 Jan 29. PMID 28128670
- [Background] Moignet A, Lamy T. Latest Advances in the Diagnosis and Treatment of Large Granular Lymphocytic Leukemia. Am Soc Clin Oncol Educ Book. 2018 May 23;38:616-625. doi: 10.1200/EDBK_200689. PMID 30231346
- [Background] Zambello R, Teramo A, Gattazzo C, Semenzato G. Are T-LGL Leukemia and NK-Chronic Lymphoproliferative Disorder really two distinct diseases? Transl Med UniSa. 2014 Feb 4;8:4-11. eCollection 2014 Jan. PMID 24778993
- [Background] Cheon H, Dziewulska KH, Moosic KB, Olson KC, Gru AA, Feith DJ, Loughran TP Jr. Advances in the Diagnosis and Treatment of Large Granular Lymphocytic Leukemia. Curr Hematol Malig Rep. 2020 Apr;15(2):103-112. doi: 10.1007/s11899-020-00565-6. PMID 32062772
- [Background] Lamy T, Moignet A, Loughran TP Jr. LGL leukemia: from pathogenesis to treatment. Blood. 2017 Mar 2;129(9):1082-1094. doi: 10.1182/blood-2016-08-692590. Epub 2017 Jan 23. PMID 28115367
- [Derived] Yu Y, Li Y, Cui R, Yan Y, Li F, Chen Y, Wang T, Hu X, Feng Y, Yu T, Huang Y, Sun J, Lyu R, Xiong W, Wang Q, Liu W, An G, Sui W, Xu Y, Huang W, Zou D, Wang H, Xiao Z, Wang J, Qiu L, Yi S. Thalidomide-based regimen shows promising efficacy in large granular lymphocytic leukemia: a multicenter phase II study. Signal Transduct Target Ther. 2025 Mar 12;10(1):85. doi: 10.1038/s41392-025-02164-4. PMID 40069155